CLINICAL TRIAL: NCT01043913
Title: Guaraná ("Paullinia Cupana") for Chemotherapy Related Fatigue in Breast Cancer Patients: Results Of A Pilot Double Blind Randomized Study
Brief Title: Guarana (Paullinia Cupana) for Breast Cancer Chemotherapy-related Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Auro Del Giglio, MD, PhD, ABC Foundation School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: mairapaschoin
Record Dates: First submitted 2009-12-22; First posted 2010-01-07 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-11

CONDITIONS: Signs and Symptoms; Neoplasms; Neoplasms by Site; Fatigue; Breast Neoplasms; Breast Diseases
Keywords: Fatigue; Breast Neoplasms; Quality of Life; Paullinia
MeSH Terms: conditions — Signs and Symptoms; Neoplasms; Neoplasms by Site; Fatigue; Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guaraná extract 50mg q12 hours (Experimental): Guaraná extract pills of 50mg q12 hours for 21 days
  Interventions: Drug: Guarana extract
- Placebo 1 tab q12 hours (Placebo Comparator): Placebo pills 1 tab q12 hours for 21 days
  Interventions: Drug: Guarana extract

INTERVENTIONS:
Drug: Guarana extract — Guarana extract 50mg q12 hours for 21 days
  Other Names: Paullinia Cupana

SUMMARY:
The investigators hypothesize that Guaraná, a native plant from the Amazon, might improve chemotherapy-induced fatigue in breast cancer patients undergoing treatment. In order to assess this, the investigators randomized patients to either guaraná extract or to placebo, switching the assigned treatment mid-term through the cycles of Chemotherapy.

DETAILED DESCRIPTION:
The aim of this study is evaluate the favourable effects of Guaraná in quality of life and Fatigue in patients undergoing Chemotherapy treatment for Breast Cancer. After approval by our Institutional Review Board, we included consenting patients with a histological diagnosis of Breast Cancer for whom Chemotherapy was indicated.

Patients who agreed to participate in the study were submitted initially to a screening interview with the Brief Fatigue Inventory questionnaire from MD Anderson. If the patient presented with a severe fatigue, anemia (HB<11.0), hypothyroidism or psychiatric disorders she was excluded. If she presented with a mild or moderate fatigue the follow up continued and the patient was assessed 21 days later after her first cycle of chemotherapy with the same questionnaire. If an increase in fatigue levels occurred from mild to moderate, mild to severe or moderate to severe the patient was randomly assigned to receive either Guaraná 50mg or a placebo p.o. q12 for 21 days. At this moment the patient answered a General questionnaire, FACIT-F, FACIT-ES, HADS, Pittsburgh Sleep Quality Index and Chalder Fatigue Questionnaire (Day 1).

After the second cycle of chemotherapy the patient underwent a "wash out" period of 7 days without any intervention, and after that period she received placebo or Guaraná according to the cross over design after answering for the second time the questionnaires above (Day 29) and also the Common Terminology Criteria for Adverse Events v3.0 (CTCAE). After 21 days (Day 42) she was assessed again with the same questionnaires used in the second interview.

The patient's cancer diagnosis, treatment history, concurrent medication was recorded during the pretreatment and The Brief Fatigue Inventory was answered before each assessment.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of Breast Cancer
* Patients undergoing Chemotherapy (First Cycle)
* 18 years old or older

Exclusion Criteria:

* Hypothyroidism
* Clinical Depression
* Prior Chemotherapy
* Anemia
* Unable to sign informed consent
* Severe Fatigue

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Fatigue improvement between the baseline to D21 or from D21 to D42 measured by Chalder Fatigue Scale, FACT-F and FACT-ES questionnaires | 42 days

SECONDARY OUTCOMES:
To access the quality of life between the baseline to D21 or from D21 to D42 measured by FACT-F and FACT ES questionnaires | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Auro D Giglio, MD, PhD, Study Director — Faculdade de Medicina do ABC; Maira P Oliveira Campos, MD, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil

REFERENCES:
- [Background] de Souza Fede AB, Bensi CG, Trufelli DC, de Oliveira Campos MP, Pecoroni PG, Ranzatti RP, Kaliks R, Del Giglio A. Multivitamins do not improve radiation therapy-related fatigue: results of a double-blind randomized crossover trial. Am J Clin Oncol. 2007 Aug;30(4):432-6. doi: 10.1097/COC.0b013e31804b40d9. PMID 17762445
- [Result] da Costa Miranda V, Trufelli DC, Santos J, Campos MP, Nobuo M, da Costa Miranda M, Schlinder F, Riechelmann R, del Giglio A. Effectiveness of guarana (Paullinia cupana) for postradiation fatigue and depression: results of a pilot double-blind randomized study. J Altern Complement Med. 2009 Apr;15(4):431-3. doi: 10.1089/acm.2008.0324. PMID 19388866
- [Result] Kennedy DO, Haskell CF, Robertson B, Reay J, Brewster-Maund C, Luedemann J, Maggini S, Ruf M, Zangara A, Scholey AB. Improved cognitive performance and mental fatigue following a multi-vitamin and mineral supplement with added guarana (Paullinia cupana). Appetite. 2008 Mar-May;50(2-3):506-13. doi: 10.1016/j.appet.2007.10.007. Epub 2007 Oct 30. PMID 18077056